CLINICAL TRIAL: NCT02601950
Title: A Phase II, Multicenter Study of the EZH2 Inhibitor Tazemetostat in Adult Subjects With INI1-Negative Tumors or Relapsed/Refractory Synovial Sarcoma
Brief Title: A Study of Tazemetostat in Adult Participants With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-202; 2015-002469-41 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-11-11 (Estimated); Results first posted 2025-03-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Malignant Rhabdoid Tumors (MRT); Rhabdoid Tumors of the Kidney (RTK); Atypical Teratoid Rhabdoid Tumors (ATRT); Selected Tumors With Rhabdoid Features; Synovial Sarcoma; INI1-negative Tumors; Malignant Rhabdoid Tumor of Ovary; Renal Medullary Carcinoma; Epithelioid Sarcoma; Poorly Differentiated Chordoma (or Other Chordoma With Sponsor Approval); Any Solid Tumor With an EZH2 GOF Mutation
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label Tazemetostat (Experimental): All cohorts will receive 800 mg oral Tazemetostat twice a day in continuous 28-day cycles.
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat (EPZ-6438) is a selective small molecule inhibitor of the histone-lysine methyltransferase EZH2 gene
  Other Names: EPZ-6438; E7438; IPN60200

SUMMARY:
This study will include participants with various types of cancer known as soft-tissue sarcomas.

Tissues that can be affected by soft tissue sarcomas include fat, muscle, blood vessels, deep skin tissues, tendons and ligaments.

Soft tissue cancers are rare and can occur almost anywhere in the body.

Part 1 of this trial will study the safety and the level that adverse effects of the study drug tazemetostat in combination with doxorubicin (current front line treatment) can be tolerated (known as tolerability).

It is also designed to establish a recommended study drug dosage for the next part of the study.

Part 2 will evaluate and compare how long participants live without their disease getting worse when receiving the study drug plus doxorubicin versus doxorubicin plus placebo (dummy treatment).

DETAILED DESCRIPTION:
This is a Phase II, multicenter, open-label, single arm, 2-stage study of tazemetostat 800 mg BID (twice daily) and 1600 mg QD (once daily). Subjects will be screened for eligibility within 21 days of the planned date of the first dose of tazemetostat and enrolled into one of 8 cohorts:

Cohort using tazemetostat 800 mg BID

* Cohort 1 (Closed for enrollment): malignant rhabdoid tumor (MRT), rhabdoid tumor of the kidney (RTK), atypical teratoid rhabdoid tumor (ATRT), and selected tumors with rhabdoid features, including small cell carcinoma of the ovary hypercalcemic type (SCCOHT), also known as malignant rhaboid tumor of the ovary (MRTO)
* Cohort 2 (Closed for enrollment): Relapsed or refractory synovial sarcoma with SS18-SSX rearrangement
* Cohort 3 (Closed for enrollment): Other integrase interactor 1 (INI1) negative tumors or any solid tumor with an enhancer of zeste homologue-2 (EZH2) gain of function (GOF) mutation, including: epithelioid malignant peripheral nerve sheath tumor (EMPNST), extraskeletal myxoid chondrosarcoma (EMC), myoepithelial carcinoma, other INI1-negative malignant tumors with Sponsor approval (e.g., dedifferentiated chordoma) any solid tumor with an EZH2 GOF mutation including but not limited to Ewing's sarcoma and melanoma
* Cohort 4 (Closed for enrollment): Renal medullary carcinoma (RMC)
* Cohort 5 (Closed for enrollment): Epithelioid sarcoma (ES)
* Cohort 6 (Closed for enrollment): Epithelioid sarcoma (ES) undergoing mandatory tumor biopsy
* Cohort 7 (Closed for enrollment): Poorly differentiated chordoma (or other chordoma with Sponsor approval)

Cohort using tazemetostat 1600 mg QD

• Cohort 8 (Closed for enrollment): Epitheliod sarcoma

Participants will be dosed in continuous 28-day cycles. (Note: if treatment with study drug is discontinued prior to completing 2 years, subjects will be followed for a maximum duration of 2 years from start of study drug dosing.) Response assessment will be performed every 8 weeks while on study.

Treatment with tazemetostat will continue until disease progression, unacceptable toxicity or withdrawal of consent, or termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age (at the time of consent/assent): ≥18 years of age
2. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
3. Has provided signed written informed consent
4. Has a life expectancy of >3 months
5. Has a malignancy:

   * For which there are no standard therapies available (Cohorts 1, 3, 4 and 5)
   * That is relapsed or refractory after treatment with an approved therapy(ies), defined as metastatic or non-resectable, locally advanced disease that has previously been treated with and progressed following approved therapy(ies) (Cohort 2)

     * That has progressed within 6 months prior to study enrollment (Cohort 5 Expansion, Cohort 6 and Cohort 8 ONLY)
6. Has a documented local diagnostic pathology of original biopsy confirmed by a Clinical Laboratory Improvement Amendments (CLIA/College of American Pathologists (CAP) or equivalent laboratory certification
7. For Cohort 1 (rhabdoid tumors only), the following test results must be available by local laboratory: morphology and immunophenotypic panel consistent with rhabdoid tumors, and loss of INI1 or SMARCA4 confirmed by IHC, or molecular confirmation of tumor bi-allelic INI1 or SMARCA4 loss or mutation when INI1 or SMARCA4 IHC is equivocal or unavailable
8. For Cohort 2 (subjects with relapsed/refractory synovial sarcoma only), the following tests must be available by local laboratory: Morphology consistent with synovial sarcomas, and cytogenetics or fluorescence in situ hybridization (FISH) and/or molecular confirmation (e.g., DNA sequencing) of SS18 rearrangement t(X;18)(p11;q11)
9. For Cohort 3, 4, 5, 7 and 8 (subjects with INI1-negative/aberrant tumors or any solid tumor with EZH2 GOF mutation only), the following test results must be available by local laboratory: Morphology and immunophenotypic panel consistent with INI1-negative tumors (not applicable for solid tumors with EZH2 GOF mutation), and loss of INI1 confirmed by IHC, or molecular confirmation of tumor bi-allelic INI1 loss or mutation when INI1 IHC is equivocal or unavailable, or molecular evidence of EZH2 GOF mutation
10. For Cohort 6 (subjects with ES undergoing optional tumor biopsy) only:

    * Morphology and immunophenotypic panel consistent with ES (e.g., CD34, EMA, Keratin, and INI1)
11. Has all prior treatment (i.e. chemotherapy, immunotherapy, radiotherapy) related clinically significant toxicities resolve to ≤Grade 1 per CTCAE version 4.0.3 or are clinically stable and not clinically significant, at time of enrollment.
12. Prior anti-cancer therapy(ies), if applicable, must be completed according to the criteria below:

    * Chemotherapy: cytotoxic (At least 14 days since last dose of chemotherapy prior to first dose of tazemetostat)
    * Chemotherapy: nitrosoureas (At least 6 weeks since last dose of nitrosoureas prior to first dose of tazemetostat)
    * Chemotherapy: non-cytotoxic (e.g., small molecule inhibitor) (At least 14 days since last dose of non-cytotoxic chemotherapy prior to first dose of tazemetostat)
    * Monoclonal antibody(ies) (At least 28 days since the last dose of any monoclonal antibody prior to first dose of tazemetostat)
    * Immunotherapy (e.g. tumor vaccine) (At least 42 days since last dose of immunotherapy agent(s) prior to first dose of tazemetostat)
    * Radiotherapy (RT) (At least 14 days from last local site RT prior to first dose of tazemetostat/At least 21 days from stereostatic radiosurgery prior to first dose of tazemetostat/At least 12 weeks from craniospinal, ≥50% radiation of pelvis, or total body irradiation prior to first dose of tazemetostat)
    * High dose therapy with autologous hematopoietic cell infusion (At least 60 days from last infusion prior to first dose of tazemetostat)
    * Hematopoietic growth factor (At least 14 days from last dose of hematopoietic growth factor prior to first dose of tazemetostat)
13. Has sufficient tumor tissue (slides or blocks) available for central confirmatory testing
14. Has measurable disease based on either RECIST 1.1 for solid tumors or RANO for CNS tumors
15. Has adequate hematologic (bone marrow [BM] and coagulation factors), renal and hepatic function.
16. For subjects with CNS Tumors only, subject must have seizures that are stable, not increasing in frequency or severity and controlled on current anti-seizure medication(s) for a minimum of 21 days prior to the planned first dose of tazemetostat
17. Has a shortening fraction of >27% or an ejection fraction of ≥50% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan and New York Heart Association (NYHA) Class ≤2
18. Has a QT interval corrected by Fridericia's formula (QTcF) ≤480 msec
19. Female subjects of childbearing potential must:

    * Have a negative beta-human chorionic gonadotropin (β-hCG) pregnancy test at time of screening and within 14 days prior to planned first dose of tazemetostat and
    * Agree to use effective contraception from a minimum of 7 days prior to first dose until 6 months following the last dose of tazemetostat and have a male partner who uses a condom, or
    * Practice true abstinence or have a male partner who is vasectomized
20. Male subjects with a female partner of childbearing potential must:

    * Be vasectomized, or
    * Agree to use condoms as defined in Section 8.6.2, from first dose of tazemetostat until 3 months following the last dose of tazemetostat, or
    * Have a female partner who is NOT of childbearing potential

Exclusion Criteria:

1. Has had prior exposure to tazemetostat or other inhibitor(s) of enhancer of zeste homologue-2 (EZH2)
2. Has participated in another interventional clinical study and received investigational drug within 30 days or 5 half-lives, whichever is longer, prior to the planned first dose of tazemetostat
3. Has known active CNS or any leptomeningeal metastasis of primary extra-cranial tumor.
4. Has had a prior malignancy other than the malignancies under study - EXCEPTION: A subject who has been disease-free for 5 years, or a subject with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma is eligible
5. Has had major surgery within 3 weeks prior to enrollment
6. Has Thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE 4.03 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS). Has abnormalities known to be associated with MDS (e.g. del 5q, chr 7 abn) and MPN (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing.
7. Has a prior history of T-LBL /T-ALL
8. Is unwilling to exclude grapefruit juice, Seville oranges and grapefruit from the diet
9. Has cardiovascular impairment, history of congestive heart failure greater than NYHA Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months prior to the planned first dose of tazemetostat; or ventricular cardiac arrhythmia requiring medical treatment
10. Is currently taking any prohibited medication(s)
11. Has an active infection requiring systemic treatment
12. Is immunocompromised (i.e. has congenital immunodeficiency), including subjects known history of infection with human immunodeficiency virus (HIV)
13. Has known active infection with hepatitis B virus or hepatitis C virus
14. Has had a symptomatic venous thrombosis within 2 weeks prior to study enrollment -
15. For subjects with CNS involvement (primary tumor or metastatic disease), have any active bleeding or new intratumoral hemorrhage of more than punctuate size of screening MRI obtained within 14 days of starting study drug or known bleeding diathesis or treatment with anti-platelet or anti-thrombotic agents
16. Has known hypersensitivity to any of the component of tazemetostat or other inhibitor(s)of EZH2
17. Is unable to take oral medications, or has a malabsorption syndrome or any uncontrolled gastrointestinal condition (e.g., nausea, diarrhea or vomiting) that would limit compliance with study requirements.
18. Has an uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements.
19. For female subjects of childbearing potential: Is pregnant or nursing
20. For male subjects: Is unwilling to adhere to contraception criteria from time of enrollment in the study to at least 3 months after last dose of tazemetostat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (32):
- United States (14):
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital - Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Metro South Hospital and Health Service via Princess Alexandra Hospital, Woolloongabba
- Belgium (2):
  - Institut Jules Bordet Medical Oncology Clinic, Brussels
  - University Hospital Leuven, Leuven
- Canada (3):
  - Alberta Health Services, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Hospital Pitie Salpetriere, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Children's Hospital Augsburg Klinikum, Augsburg
  - Sarcoma Center HELIOS Klinikum Berlin, Berlin
- Instituto Nazionale Tumori - National Cancer Institute Via Giacomo Venezian, Milan, Italy
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (2):
  - University College London Hospital, London
  - Royal Marsden Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Gounder M, Schoffski P, Jones RL, Agulnik M, Cote GM, Villalobos VM, Attia S, Chugh R, Chen TW, Jahan T, Loggers ET, Gupta A, Italiano A, Demetri GD, Ratan R, Davis LE, Mir O, Dileo P, Van Tine BA, Pressey JG, Lingaraj T, Rajarethinam A, Sierra L, Agarwal S, Stacchiotti S. Tazemetostat in advanced epithelioid sarcoma with loss of INI1/SMARCB1: an international, open-label, phase 2 basket study. Lancet Oncol. 2020 Nov;21(11):1423-1432. doi: 10.1016/S1470-2045(20)30451-4. Epub 2020 Oct 6. PMID 33035459
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2025/02/26115902/ezh202-lay-results-summary-EN.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II, open-label study was conducted at 28 sites in 9 countries (Australia, Belgium, Canada, France, Germany, Italy, Taiwan, United Kingdom, and United States) from 22 December 2015 to 26 February 2024.
Pre-assignment Details: Participants were enrolled into 1 of the 8 cohorts based on tumor type. A total of 267 participants were enrolled in the study.
Groups:
- Rhabdoid Tumors: Cohort 1: Participants with rhabdoid tumors (malignant rhabdoid tumor [MRT], rhabdoid tumors of the kidney [RTK], atypical teratoid rhabdoid tumor [ATRT], and selected tumors with rhabdoid features, including small cell carcinoma of the ovary hypercalcemic type [SCCOHT], also known as malignant rhabdoid tumor of the ovary [MRTO]) received tazemetostat 800 milligram (mg) twice daily (BID) orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- Synovial Sarcoma: Cohort 2: Participants with relapsed or refractory synovial sarcoma with SS18-SSX rearrangement received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- Other INI1-negative: Cohort 3: Participants with other integrase interactor 1 (INI-1)-negative tumors or any solid tumor with enhancer of zeste homologue-2 (EZH2) gain of function (GOF) mutation, including epithelioid malignant peripheral nerve sheath tumor (EMPNST), extraskeletal myxoid chondrosarcoma (EMC), myoepithelial carcinoma, other INI-1-negative malignant tumors with sponsor approval, any solid tumor with EZH2 GOF mutation including but not limited to Ewing's sarcoma and melanoma received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- RMC: Cohort 4: Participants with renal medullary carcinoma (RMC) received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- ES: Cohort 5: Participants with epithelioid sarcoma (ES) received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- ES Paired Biopsy: Cohort 6: Participants with ES undergoing optional tumor biopsy received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- Chordoma: Cohort 7: Participants with poorly differentiated chordoma (or other chordoma with sponsor approval) received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- ES 1600 mg: Cohort 8: Participants with ES received tazemetostat 1600 mg once daily (QD) orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
Period: Overall Study
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
Started | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7
Not completed — Participant enrolled in rollover study | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Disease progression - radiological | 21 | 26 | 22 | 11 | 46 | 52 | 7 | 5
Not completed — Disease progression - clinical | 3 | 5 | 4 | 2 | 6 | 6 | 5 | 1
Not completed — Death | 6 | 0 | 3 | 1 | 4 | 1 | 0 | 0
Not completed — Unacceptable toxicity (related to study treatment) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse event (not related to study treatment) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Participant refused further study treatment | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 1
Not completed — Investigator discretion | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of tazemetostat.
Groups:
- Rhabdoid Tumors: Cohort 1: Participants with rhabdoid tumors (MRT, RTK, ATRT, and selected tumors with rhabdoid features, including SCCOHT, also known as MRTO) received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- Other INI1-negative: Cohort 3: Participants with other INI-1-negative tumors or any solid tumor with EZH2 GOF mutation, including EMPNST, EMC, myoepithelial carcinoma, other INI-1-negative malignant tumors with sponsor approval, any solid tumor with EZH2 GOF mutation including but not limited to Ewing's sarcoma and melanoma received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- RMC: Cohort 4: Participants with RMC received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- ES: Cohort 5: Participants with ES received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- ES Paired Biopsy: Cohort 6: Participants with ES undergoing optional tumour biopsy received tazemetostat 800 mg BID orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- ES 1600 mg: Cohort 8: Participants with ES received tazemetostat 1600 mg QD orally in continuous 28-day cycles until disease progression, development of an unacceptable toxicity, withdrawal of consent, or termination of the study.
- Total: Total of all reporting groups
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8 | Total
Number analyzed (Participants) | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (16.31) | 38.8 (9.54) | 46.9 (16.94) | 30.7 (10.71) | 37.0 (15.08) | 41.3 (14.00) | 38.9 (17.49) | 40.9 (15.74) | 39.5 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 17 | 4 | 23 | 26 | 8 | 4 | 113
  Male | 13 | 21 | 15 | 10 | 39 | 43 | 10 | 3 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 4 | 1 | 7 | 4 | 0 | 0 | 21
  Not Hispanic or Latino | 31 | 28 | 27 | 13 | 53 | 55 | 17 | 7 | 231
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2 | 10 | 1 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 1 | 0 | 7 | 9 | 1 | 2 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 4 | 2 | 11 | 4 | 1 | 1 | 0 | 26
  White | 24 | 24 | 28 | 2 | 47 | 54 | 16 | 5 | 200
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 1 | 1 | 4 | 4 | 0 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1, 3, 4, 5, 6 and 7: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants who achieved a confirmed complete response (CR) or partial response (PR) based on the investigator review from start of treatment until progressive disease (PD) or start of subsequent anti-cancer therapy or cancer-related surgery, whichever was earlier, as per response assessment in neuro-oncology (RANO) criteria for primary brain tumors or response evaluation criteria in solid tumors (RECIST) version (v) 1.1 criteria for all other solid tumors. CR was defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must be <10 millimeter (mm) in short axis. PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as a reference, baseline sum of diameters. PD was defined as at least a 20% increase in sum of diameters of target lesions, taking as a reference, smallest sum of diameters recorded since treatment started. In addition, sum must have an absolute increase from nadir of 5 mm.
Time Frame: Tumor assessment performed at screening and every 8 weeks beginning at Cycle 3 Day 1, until disease progression or the start of subsequent anti-cancer therapy, whichever occurred first, up to 5.75 years (cycle duration: 28 days)
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rhabdoid Tumors: Cohort 1 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7
Number analyzed (Participants) | 32 | 32 | 14 | 62 | 69 | 18
Percentage of participants | 9.4 [2.0 to 25.0] | 9.4 [2.0 to 25.0] | 0.0 [0.0 to 23.2] | 16.1 [8.0 to 27.7] | 15.9 [8.2 to 26.7] | 5.6 [0.1 to 27.3]

2. Primary Outcome: Cohort 2: Progression-Free Survival (PFS) Rate at 16 Weeks of Treatment With Tazemetostat
Description: PFS was defined as the interval of time between the date of the first dose of study treatment and the earliest date of PD or death due to any cause, whichever comes first, as per RECIST v 1.1 criteria. PFS rate at 16 week was estimated. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as a reference, smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: At 16 Weeks
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Synovial Sarcoma: Cohort 2
Number analyzed (Participants) | 33
Percentage of participants | 15.2 [5.1 to 31.9]

3. Primary Outcome: Cohort 8: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect or was medically significant. TEAEs were defined as AEs if one of the following conditions met: emerged after the time of first dose administration, having been absent prior to the first dose; re-emerged, having been present but stopped prior to the time of first dose administration; worsened in severity after the time of first dose administration relative to the pretreatment state, when the AE was continuous.
Time Frame: From first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 148 weeks
Population: Safety population included all participants in the ITT population who had at least 1 post-dose safety observation recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 7
Participants
  TEAEs | 7
  TESAEs | 2

4. Secondary Outcome: All Cohorts: Duration of Response (DOR)
Description: DOR was defined as time from the first documented evidence of CR or PR based on investigator review to the time of first documented PD or death due to any cause, whichever came first, as per RECIST v 1.1 criteria. CR was defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as a reference, baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as a reference, smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: Tumor assessment performed at screening and every 8 weeks beginning at Cycle 3 Day 1, until disease progression or the start of subsequent anti-cancer therapy, whichever occurred first, up to 5.75 years (cycle duration 28 days)
Population: ITT population included all participants who received at least 1 dose of tazemetostat. Only those participants with a confirmed CR or PR (responders) were analyzed.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 3 | 0 | 3 | 0 | 10 | 11 | 1 | 1
Weeks | 29.0 [24.1 to 32.1] |  | 80.1 [24.1 to 87.6] |  | 88.0 [7.1 to 224.4] | 96.1 [10.3 to 112.3] | 151.6 [151.6 to 151.6] | 119.4 [119.4 to 119.4]

5. Secondary Outcome: All Cohorts: Progression-Free Survival (PFS)
Description: PFS was defined as the interval of time between the date of the first dose of study treatment and the earliest date of PD or death due to any cause, whichever comes first, as per RECIST v 1.1 criteria. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as a reference, smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: as for outcome 4
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7
Weeks | 7.9 [7.7 to 15.1] | 8.0 [7.6 to 8.1] | 15.7 [7.7 to 31.7] | 7.3 [6.3 to 15.1] | 23.7 [14.7 to 25.7] | 16.1 [8.4 to 16.6] | 24.0 [6.3 to 175.3] | 39.9 [4.1 to NA] — NA indicates that upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events at study closure.

6. Secondary Outcome: All Cohorts: Progression-Free Survival (PFS) Rate at Weeks 24, 32 and 56
Description: PFS was defined as the interval of time between the date of the first dose of study treatment and the earliest date of PD or death due to any cause, whichever comes first, as per RECIST v 1.1 criteria. PFS rate at 24, 32 and 56 weeks were estimated. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as a reference, smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase from nadir of 5 mm. Estimates were calculated with Kaplan-Meier analysis and 95% CIs using the complementary log-log transformation.
Time Frame: At Weeks 24, 32 and 56
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7
Percentage of participants
  Week 24 | 17.6 [6.5 to 33.1] | 15.9 [5.1 to 32.0] | 34.4 [18.2 to 51.2] | 15.4 [2.5 to 38.8] | 42.1 [29.3 to 54.4] | 33.8 [22.9 to 45.0] | 43.6 [18.2 to 66.7] | 53.6 [13.2 to 82.5]
  Week 32 | 14.1 [4.5 to 28.9] | 10.6 [2.2 to 26.7] | 26.7 [12.3 to 43.5] | 15.4 [2.5 to 38.8] | 29.1 [17.9 to 41.2] | 29.3 [19.1 to 40.4] | 43.6 [18.2 to 66.7] | 53.6 [13.2 to 82.5]
  Week 56 | 3.5 [0.3 to 15.2] | 0.0 [0.0 to 0.0] | 13.8 [3.8 to 29.9] | 0.0 [0.0 to 0.0] | 21.3 [11.6 to 33.0] | 22.6 [13.3 to 33.3] | 18.2 [1.5 to 50.3] | 26.8 [1.3 to 67.0]

7. Secondary Outcome: All Cohorts: Overall Survival (OS)
Description: OS was defined as the interval of time between the date of the first dose of study treatment and the date of death due to any cause.
Time Frame: as for outcome 1
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7
Weeks | 22.1 [14.4 to 54.6] | 43.4 [31.7 to 58.1] | 37.9 [23.3 to 104.0] | 24.6 [8.4 to 73.6] | 82.4 [47.4 to 117.0] | 111.4 [63.0 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 77.7 [32.9 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 49.6 [19.3 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure.

8. Secondary Outcome: All Cohorts: Overall Survival (OS) Rate at Weeks 24, 32 and 56
Description: OS was defined as the interval of time between the date of the first dose of study treatment and the date of death due to any cause. OS rate at 24, 32 and 56 weeks were estimated. Estimates were calculated with Kaplan-Meier analysis and 95% CIs using the complementary log-log transformation.
Time Frame: At Weeks 24, 32 and 56
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7
Percentage of participants
  Week 24 | 45.4 [27.6 to 61.6] | 81.4 [63.2 to 91.2] | 68.8 [49.7 to 81.8] | 50.0 [22.9 to 72.2] | 85.5 [73.9 to 92.2] | 83.6 [72.3 to 90.6] | 88.9 [62.4 to 97.1] | 83.3 [27.3 to 97.5]
  Week 32 | 38.6 [21.8 to 55.2] | 68.9 [49.9 to 81.9] | 56.3 [37.6 to 71.3] | 42.9 [17.7 to 66.0] | 77.2 [64.6 to 85.8] | 75.8 [63.6 to 84.4] | 77.8 [51.1 to 91.0] | 66.7 [19.5 to 90.4]
  Week 56 | 30.9 [15.5 to 47.7] | 37.6 [21.3 to 53.8] | 49.6 [31.4 to 65.4] | 35.7 [13.0 to 59.4] | 57.3 [43.9 to 68.6] | 66.5 [53.7 to 76.6] | 55.6 [30.5 to 74.8] | 44.4 [6.6 to 78.5]

9. Secondary Outcome: All Cohorts: Disease Control Rate (DCR) at Weeks 12, 24, 32 and 48
Description: DCR was defined as the percentage of participants who achieved a confirmed response (CR or PR, as per RECIST v 1.1 criteria) or who have SD lasting at least 32 weeks from the start of treatment until disease progression or the start of subsequent anti-cancer therapy. CR was defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as a reference, baseline sum of diameters. SD was defined neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: At Weeks 12, 24, 32 and 48
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 32 | 33 | 32 | 14 | 62 | 69 | 18 | 7
Percentage of participants
  Week 12 | 21.9 [9.3 to 40.0] | 15.2 [5.1 to 31.9] | 40.6 [23.7 to 59.4] | 21.4 [4.7 to 50.8] | 45.2 [32.5 to 58.3] | 36.2 [25.0 to 48.7] | 50.0 [26.0 to 74.0] | 42.9 [9.9 to 81.6]
  Week 24 | 12.5 [3.5 to 29.0] | 9.1 [1.9 to 24.3] | 21.9 [9.3 to 40.0] | 14.3 [1.8 to 42.8] | 29.0 [18.2 to 41.9] | 30.4 [19.9 to 42.7] | 33.3 [13.3 to 59.0] | 42.9 [9.9 to 81.6]
  Week 32 | 9.4 [2.0 to 25.0] | 3.0 [0.1 to 15.8] | 18.8 [7.2 to 36.4] | 7.1 [0.2 to 33.9] | 25.8 [15.5 to 38.5] | 29.0 [18.7 to 41.2] | 27.8 [9.7 to 53.5] | 14.3 [0.4 to 57.9]
  Week 48 | 9.4 [2.0 to 25.0] | 3.0 [0.1 to 15.8] | 12.5 [3.5 to 29.0] | 0.0 [0.0 to 23.2] | 24.2 [14.2 to 36.7] | 23.2 [13.9 to 34.9] | 11.1 [1.4 to 34.7] | 14.3 [0.4 to 57.9]

10. Secondary Outcome: Cohorts 2 and 8: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants who achieved a confirmed CR or PR based on investigator assessment from start of treatment until PD or start of subsequent anti-cancer therapy or cancer-related surgery, whichever was earlier, as per RANO criteria for primary brain tumors or RECIST v 1.1 criteria for all other solid tumors. CR was defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as a reference, baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as a reference, smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: as for outcome 1
Population: ITT population included all participants who received at least 1 dose of tazemetostat.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Synovial Sarcoma: Cohort 2 | ES 1600 mg: Cohort 8
Number analyzed (Participants) | 33 | 7
Percentage of participants | 0 [0.0 to 10.6] | 14.3 [0.4 to 57.9]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 88 weeks (Cohort 1), 55 weeks (Cohort 2), 148 weeks (Cohorts 3 and 8), 48 weeks (Cohort 4), 304 weeks (Cohort 5), 270 weeks (Cohort 6) and 183 weeks (Cohort 7). All-cause mortality (deaths) were collected from first dose of study treatment (Day 1) up to 5.75 years.
Description: Safety population included all participants in the ITT population who had at least 1 post-dose safety observation recorded.
Arm/Group | Rhabdoid Tumors: Cohort 1 | Synovial Sarcoma: Cohort 2 | Other INI1-Negative: Cohort 3 | RMC: Cohort 4 | ES: Cohort 5 | ES Paired Biopsy: Cohort 6 | Chordoma: Cohort 7 | ES 1600 mg: Cohort 8
All-Cause Mortality (participants affected / at risk) | 9/32 | 2/33 | 5/32 | 3/14 | 8/62 | 6/69 | 2/18 | 0/7
Serious Adverse Events (participants affected / at risk) | 18/32 | 13/33 | 11/32 | 8/14 | 25/62 | 19/69 | 7/18 | 2/7
Other Adverse Events (participants affected / at risk) | 27/32 | 28/33 | 29/32 | 12/14 | 58/62 | 65/69 | 16/18 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rhabdoid Tumors: Cohort 1 (N=32) | Synovial Sarcoma: Cohort 2 (N=33) | Other INI1-Negative: Cohort 3 (N=32) | RMC: Cohort 4 (N=14) | ES: Cohort 5 (N=62) | ES Paired Biopsy: Cohort 6 (N=69) | Chordoma: Cohort 7 (N=18) | ES 1600 mg: Cohort 8 (N=7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (6) | 2 (2) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 1 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 0 (0) | 4 (4) | 3 (3) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2) | 2 (3) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rhabdoid Tumors: Cohort 1 (N=32) | Synovial Sarcoma: Cohort 2 (N=33) | Other INI1-Negative: Cohort 3 (N=32) | RMC: Cohort 4 (N=14) | ES: Cohort 5 (N=62) | ES Paired Biopsy: Cohort 6 (N=69) | Chordoma: Cohort 7 (N=18) | ES 1600 mg: Cohort 8 (N=7)
Nausea (Gastrointestinal disorders) | 10 (15) | 9 (14) | 9 (18) | 3 (3) | 23 (31) | 32 (43) | 8 (10) | 3 (5)
Vomiting (Gastrointestinal disorders) | 13 (18) | 1 (2) | 9 (12) | 5 (6) | 16 (23) | 9 (13) | 5 (5) | 3 (5)
Constipation (Gastrointestinal disorders) | 7 (7) | 4 (4) | 5 (5) | 4 (4) | 13 (17) | 10 (10) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 3 (3) | 6 (6) | 0 (0) | 10 (15) | 16 (17) | 3 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (3) | 1 (1) | 4 (7) | 7 (8) | 1 (1) | 1 (1)
Fatigue (General disorders) | 7 (7) | 10 (13) | 11 (12) | 3 (3) | 24 (38) | 21 (26) | 4 (6) | 3 (6)
Asthenia (General disorders) | 3 (3) | 4 (8) | 3 (3) | 0 (0) | 4 (6) | 9 (14) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 2 (2) | 1 (1) | 2 (2) | 6 (6) | 7 (8) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (8) | 5 (6) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 10 (12) | 4 (6) | 3 (3) | 13 (13) | 5 (6) | 2 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (9) | 4 (4) | 4 (4) | 6 (7) | 7 (11) | 0 (0) | 3 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (4) | 3 (3) | 4 (5) | 4 (5) | 0 (0) | 4 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1) | 6 (6) | 1 (1) | 7 (7) | 4 (6) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 4 (4) | 9 (10) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 7 (7) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 11 (11) | 3 (3) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 8 (13) | 7 (9) | 2 (3) | 19 (29) | 1 (1) | 2 (3) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 4 (7) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 3 (4) | 8 (9) | 15 (27) | 9 (9) | 3 (3) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 2 (5) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 3 (5) | 1 (1) | 11 (17) | 5 (6) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 2 (5) | 2 (3) | 4 (6) | 10 (22) | 6 (12) | 0 (0) | 3 (4)
Weight increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 6 (17) | 3 (4) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (7) | 4 (8) | 4 (6) | 4 (5) | 10 (34) | 8 (9) | 3 (3) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 5 (5) | 7 (9) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (6) | 5 (5) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4) | 3 (3) | 5 (6) | 4 (4) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 4 (15) | 0 (0) | 7 (8) | 4 (10) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 5 (12) | 1 (1) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02601950/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT02601950/SAP_001.pdf